CLINICAL TRIAL: NCT02215876
Title: A Phase II (Single Center) Study of Neoadjuvant Doxorubicin/Cyclophosphamide Followed by Eribulin Chemotherapy (ACE) in Operable HER2-negative Breast Cancer
Brief Title: Neoadjuvant Doxorubicin/Cyclophosphamide Followed by Eribulin Chemotherapy (ACE) in Operable HER2-negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients recruited.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS1405; 2013/01251 (Other: DSRB)
Record Dates: First submitted 2014-08-06; First posted 2014-08-13 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Her 2-negative breast cancer; neoadjuvant doxorubicin/cyclophosphamide followed by Eribulin chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Doxorubucin and Cyclophosphamide q2 or q3 weekly x 4 cycles plus Eribulin on days 1 and 8 of a 21 day cycle x 4 cycles
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Eribulin

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 60mg/m2 administered intravenously over 5 minutes on day 1 of a 14 of 21 days cycle IV for 4 cycles
Drug: Cyclophosphamide — Cyclophosphamide 600mg/m2 administered intravenously over 60 minutes on day 1 of a 14 of 21 days cycle IV for 4 cycles
Drug: Eribulin — Eribulin 1.4 mg/m2 administered intravenously over 2-5 minutes on days 1 and 8 of a 21 day cycle for 4 cycles

SUMMARY:
This is a phase II, single institutional study, to evaluate a novel neo-adjuvant regimen in patients with operable, HER2-negative, breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent
2. Target Population

   1. Histologically confirmed primary invasive adenocarcinoma of the breast.
   2. Patients with operable, T2-4, N0-3, M0, T1N1 breast cancer (stage IIA, IIB, IIIA, IIIB and IIIC) with minimum tumor size of 2 cm
   3. Tumors must be HER-2/neu expression negative, as determined by local hospital laboratory (IHC ≤ 2+ or FISH negative).
   4. No prior treatment (irradiation, chemotherapy, hormonal, immunotherapy or investigational, etc.) for breast cancer excluding therapy for DCIS. Subjects receiving hormone replacement therapy (HRT) are eligible if this therapy is discontinued at least 2 weeks before starting study therapy.
   5. Subjects who received radiotherapy for DCIS may enroll.
   6. Disease free of prior malignancy for ≥ 5 years with the exception of curatively treated basal cell carcinoma of the skin or carcinoma in situ of the cervix.
   7. ECOG PS of 0 or 1.
   8. Accessible for treatment and follow-up.
   9. Baseline cardiac echocardiogram scan with LVEF of ≥ 50%.
   10. Adequate recovery from recent surgery. At least one week must have elapsed from minor surgery (placement of venous access device or fine needle aspiration) and at least 4 weeks from major surgery.
3. Laboratory Parameters

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3
   2. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN).
   3. AST or ALT ≤ 2.5 times the upper limit of normal (ULN).
   4. Platelets ≥ 100,000/ mm3.
   5. Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance > 60 mL/min (measured or calculated by Cockcroft-Gault method).
   6. Normal PTT and either INR or PT < 1.5 x ULN.
4. Age and Sex Women, at least 21 years of age. a) Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the last dose of chemotherapy in such a manner that the risk of pregnancy is minimized.

WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation,or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea ≥ 12 consecutive months; or women on hormone replacement therapy [HRT] with documented serum follicle stimulating hormone [FSH] level > 35 mIU/mL). Even women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or whose partner is sterile (vasectomy) should be considered to be of childbearing potential.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the first dose of investigational product.

Exclusion Criteria:

1. Sex and Reproductive Status

   1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of chemotherapy.
   2. Women who are pregnant (including positive pregnancy test at enrollment or prior to study drug administration) or breastfeeding.
2. Target Disease Exceptions

   1. Evidence of metastatic breast cancer following a standard tumor staging work-up.
   2. Evidence of inflammatory breast cancer.
   3. Evidence of baseline sensory or motor neuropathy.
3. Medical History and Concurrent Diseases

   1. Known human immunodeficiency viral (HIV) infection.
   2. Serious intercurrent infections or non-malignant medical illnesses that are uncontrolled or the control of which may be jeopardized by this therapy.
   3. Psychiatric disorders or other conditions rendering the subject incapable of complying with the requirements of the protocol.
   4. Clinically significant history of cardiovascular disease (history of unstable angina, congestive heart failure, uncontrolled hypertension, myocardial infarction or valvular heart disease).
   5. Subjects unfit for breast and/or axillary surgery (complete fixation of tumor, skin infiltration, erythema of the breast, and/or ulceration).
   6. Current participation in another drug trial.
   7. Subjects who received prior anthracycline therapy.
   8. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical illness (e.g., infectious disease) must not be enrolled into this study.

   Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and to ensure that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.
4. Allergies and Adverse Drug Reactions

   a) Known allergy to any of the study drugs
5. Prohibited Therapies and/or Medications a) Other concurrent anti-tumor, chemotherapy, hormonal therapy, immunotherapy regimens or radiation therapy, standard or investigational.

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic Response Rate | Estimated 6 months
  To evaluate the pathologic complete response (pCR) rate following neoadjuvant treatment with four cycles of Doxorubicin and Cyclophosphamide (AC) and four cycles of Eribulin mesylate chemotherapy in HER2-negative operable breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Chopra, Principal Investigator — Johns Hopkins Singapore
Locations (1):
- Johns Hopkins Singapore, Singapore, Singapore, Singapore